CLINICAL TRIAL: NCT01468194
Title: Change in Peripheral Oxygen Saturation by Using Different Breathing Procedures in High Altitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Giessen (Other)
Collaborators: MVZ für Laboratoriumsmedizin Koblenz (Unknown)
Responsible Party: Principal Investigator, Andree Hillebrecht, Akademischer Rat, University of Giessen
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: Gi-04-2011
Record Dates: First submitted 2011-10-09; First posted 2011-11-09 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Acute Mountain Sickness
Keywords: AMS; HAPE; high altitude; oxygen; saturation; mountain; climbing; breathing
MeSH Terms: conditions — Altitude Sickness; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Breathing procedure 1 (Experimental): Walking with breathing procedure "1".
  Interventions: Other: Breathing procedure 1
- Breathing procedure 2 (Experimental): Walking with breathing procedure "2".
  Interventions: Other: Breathing procedure 2
- Control group (No Intervention): Walking without any reglementation of breathing

INTERVENTIONS:
Other: Breathing procedure 1 — inhalation during one step, exhalation during the next step
  Arms: Breathing procedure 1
Other: Breathing procedure 2 — inhalation and exhalation during one step
  Arms: Breathing procedure 2

SUMMARY:
In this investigation the researchers explore whether different types of breathing procedures can improve the peripheral oxygen saturation to reduce the risk of becoming a acute mountain sickness or a high altitude pulmonary edema.

DETAILED DESCRIPTION:
Acute mountain sickness (AMS) is a pathological effect of high altitude on humans caused by acute exposure to low partial pressure of oxygen at high altitude. It commonly occurs above 2500 meters of altitude. AMS appears as a collection of nonspecific symptoms acquired at high altitude or in low air pressure resembling a case of "flu, carbon monoxide poisoning, or a hangover".

It is caused by a drop in pressure and lowering partial pressure of oxygen during increasing altitude. The direct consequence of those changes is a hypoxic pulmonary vasoconstriction (Euler-Lijestrand-mechanism). In addition a rise in pulmonary blood pressure (Hypertonia) can occur so that there is a higher risk of developing a high altitude pulmonary edema (HAPE).

In this investigation the investigators are exploring whether different types of breathing procedures can improve the peripheral oxygen saturation. We are comparing breathing with no regulation with two different procedures of hyperventilation during trekking in different altitudes. Procedure 1 (hyperventilation 1) describes inhalation during one step and exhalation during the next step. Procedure 2 (hyperventilation 2) describes inhalation and exhalation during one step.

The effect of the different breathing procedures can be quantified measuring the peripheral oxygen saturation. In addition the investigators are comparing the breathing rate and the minute ventilation as well as the expiratory end-tidal CO2-partial pressure of the three different breathing procedures.

Furthermore, the investigators are examining the ability to concentrate in order to quantify the effect of AMS on organ functions.

ELIGIBILITY:
Exclusion Criteria:

* acute clinically significant inter-current diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
change of peripheral oxygen saturation | immediate after intervention
  change of peripheral oxygen saturation under different breathing procedures in different altitudes

SECONDARY OUTCOMES:
change of breathing parameters | immediate after intervention
  change of breathing parameters under different breathing procedures in different altitudes
  * breathing rate
  * minute ventilation
  * expiratory end-tidal CO2-partial pressure
change of cognition | immediate after intervention
  change of ability of cognition (measured by d2-test) under different breathing procedures in different altitudes

CONTACTS AND LOCATIONS:
Overall Officials: Gabor Szalay, Dr. med., Principal Investigator — Trauma surgery - University hospital Giessen
Locations (1):
- University of Giessen, Giessen, Hesse, Germany